CLINICAL TRIAL: NCT03185715
Title: Single or Double Embryo Transfer? Decision-making Process in Patients Participating in an Oocyte Donation Program
Brief Title: Oocyte Recipient's Decision in the Number of Embryos to be Transferred
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Elisabet Clua Obrado, PhD, Fundacion Dexeus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SMD-2014-121
Record Dates: First submitted 2017-05-19; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Decision Making; Infertility, Female; Counseling
Keywords: oocyte donation; recipient counselling; single embryo transfer (SET); double embryo transfer (DET); decision-making
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Counseling policy embryo transfer (Other): All recipients completed a validated self-report questionnaire on the preference on the number of embryos to be transferred and the relevance for the decision-making process attributed to certain factors. The questionnaire also included questions on sociodemographic characteristics, medical-reproductive background and cycle's results and risks perception. All recipients received oral and written counselling. After counselling, during the treatment, the recipients completed a second questionnaire in order to check if their decision had changed.
  Interventions: Behavioral: Oral and written counselling

INTERVENTIONS:
Behavioral: Oral and written counselling — Recipients were informed about success rates of SET and DET and also about the possible risks of DET. All the information was given orally and written.

SUMMARY:
Multiple pregnancies are considered an ART complication. The only effective way to reduce its incidence is to transfer a single embryo. Nonetheless, there is some reluctance among the patients to accept this strategy. In IVF/ICSI programs, it has been demonstrated that, after receiving the information about the similar cumulative live birth rate after single embryo transfer (SET) and double embryo transfer (DET) and the obstetric and perinatal risks of multiple pregnancy, a significant number of patients opt for SET. Up to date, no comparable studies have been published in oocyte recipients. The aim of this study is to evaluate if the information given to the patients influence their preference on the number of embryos to be transferred. It also seeks to identify factors which determine the initial preference and factors which can explain a hypothetic change in this preference.

ELIGIBILITY:
Inclusion Criteria:

* Patients under their first oocyte or embryo donation cycle.
* Sufficient knowledge of Spanish to fill out questionnaires.

Exclusion Criteria:

* Patients with a medical indication for single embryo transfer (e.g. Turner syndrome, uterine surgeries, cardiovascular risk).
* Having had previous oocyte or embryo donation cycles.
* Insufficient knowledge of Spanish.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Preference change on the number of embryos to be transferred | Up to 3 months
  Preference was evaluated at the first consultation and after counselling using a self-report questionnaire.

SECONDARY OUTCOMES:
Factors which determine the initial preference on the number of embryos to be transferred | At the first consultation
  Factor's weight is analysed using a self-report questionnaire. Each factor is scored 1-10 according its relevance.
Factors which can explain a change in the preference on the number of embryos to be transferred | Up to 3 months
  Each factor is scored 1-10 according its relevance. Score before counselling and score after counselling were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Clua, PhD, Principal Investigator — Fundacion Dexeus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Land JA, Evers JL. Risks and complications in assisted reproduction techniques: Report of an ESHRE consensus meeting. Hum Reprod. 2003 Feb;18(2):455-7. doi: 10.1093/humrep/deg081. PMID 12571190
- [Background] van Peperstraten AM, Nelen WL, Hermens RP, Jansen L, Scheenjes E, Braat DD, Grol RP, Kremer JA. Why don't we perform elective single embryo transfer? A qualitative study among IVF patients and professionals. Hum Reprod. 2008 Sep;23(9):2036-42. doi: 10.1093/humrep/den156. Epub 2008 Jun 18. PMID 18565969
- [Background] Ryan GL, Sparks AE, Sipe CS, Syrop CH, Dokras A, Van Voorhis BJ. A mandatory single blastocyst transfer policy with educational campaign in a United States IVF program reduces multiple gestation rates without sacrificing pregnancy rates. Fertil Steril. 2007 Aug;88(2):354-60. doi: 10.1016/j.fertnstert.2007.03.001. Epub 2007 May 9. PMID 17490657
- [Background] Hope N, Rombauts L. Can an educational DVD improve the acceptability of elective single embryo transfer? A randomized controlled study. Fertil Steril. 2010 Jul;94(2):489-95. doi: 10.1016/j.fertnstert.2009.03.080. Epub 2009 May 13. PMID 19442970